CLINICAL TRIAL: NCT04932551
Title: Perspectives and Management of Atypical Asthma in Chinese Specialists and Primary Care Practitioners -- A Nationwide Questionnaire Survey.
Brief Title: Perspectives and Management of Atypical Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0372
Record Dates: First submitted 2021-06-03; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physician
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — physicians will participate in the questionnaire via WeChat. The questionnaire included six main items: physician demographic characteristics, awareness, diagnosis, medical prescription, assessment/education, and proposal.

SUMMARY:
To evaluate the awareness/knowledge, clinical practice of atypical asthma among respiratory specialists and primary care practitioners (PCPs) in China.A total of 1166 respiratory specialists and 799 PCPs participated in the questionnaire survey via WeChat. The questionnaire included six major items, divided into physician demographic characteristics, awareness, diagnosis, medication prescription, assessment/education, and proposal.

ELIGIBILITY:
Inclusion Criteria:

* Grade Hospital Respiratory Doctor，Pediatrician，And doctors in primary hospitals

Exclusion Criteria:

* none

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physician
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete the questionnaire | 30 minutes
  The questionnaire included six main items: physician demographic characteristics, awareness, diagnosis, medical prescription, assessment/education, and proposal.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China